CLINICAL TRIAL: NCT05295173
Title: A Phase III, Multicenter, Randomized, Blind Endpoint and Positive Drug Control Study of Recombinant Human Tissue Plasminogen Kinase Derivatives for Injection in the Treatment of Patients With Acute Ischemic Stroke
Brief Title: A Study of r-PA Treating Patients With Acute Ischemic Stroke（RAISE）
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Angde Biotech Pharmaceutical Co., Ltd. (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD-001-03
Record Dates: First submitted 2022-02-24; First posted 2022-03-25 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — reteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Recombinant human tissue plasminogen kinase derivatives(r-PA) for injection: the first intravenous bolus injection of 18mg, after 30mins, the second intravenous bolus injection of 18 mg, Push slowly for more than 2mins each time. Subjects were closely monitored during the treatment period and within 24 hours after administration.
  Interventions: Drug: Injection of recombinant human tissue plasminogen kinase derivatives
- comparative group (Active Comparator): Recombinant human tissue plasminogen activator (rt-PA) for injection: 0.9 mg/kg (maximum dose of 90 mg) intravenous, 10% of which was injected intravenously within the first 1min, and the rest continued intravenous infusion for 1 h. Subjects should be closely monitored during the treatment period and within 24 hours after administration.
  Interventions: Drug: Recombinant human tissue plasminogen activator

INTERVENTIONS:
Drug: Injection of recombinant human tissue plasminogen kinase derivatives — 18mg/10ml/stick, provided by Angde Biotech
  Other Names: Reteplase; brand name: Ruitongli; r-PA
  Arms: experimental group
Drug: Recombinant human tissue plasminogen activator — 20mg/stick, 50mg/stick, provided by Shanghai Boehringer Ingelheim Pharmaceutical Co. Ltd.
  Other Names: Alteplase; brand name: Actilyse; rt-PA
  Arms: comparative group

SUMMARY:
The purpose of this study is to assess the efficacy and safety of recombinant human tissue plasminogen kinase derivatives for injection and alteplase in the treatment of patients with acute ischemic stroke within 4.5 hours.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, blind endpoint and positive drug control study.

The study plans to recruit 1412 AIS patients within 4.5 hours of onset. Qualified subjects are assigned to the test drug and control drug alteplase group according to the ratio of 1:1. After receiving thrombolytic drugs, the subjects need to carry out a series of safety and effectiveness tests. The mRS score and Barthel index score visits are carried out on the 90th day (± 7 days) after thrombolysis. After the visit, the subjects can leave the group.

In this study, independent blind endpoint evaluators were set up in each research center to evaluate the mRS and Barthel index score 30 and 90 days after thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years（including the critical value);
2. Acute ischemic stroke is diagnosed according to the WHO (World Health Organization) stroke diagnostic criteria, the symptoms of acute ischemic stroke are expected to be less than 4.5 hours after the time of acute ischemic stroke which is defined as the last time the patient functions well;
3. NIHSS score at the time of treatment: from 4 points to 25 points (including 4 points and 25 points);
4. From the signing of informed consent form to 3 months after treatment, fertile men and women of childbearing age should be absent of a birth plan and willing to take effective contraceptive measures;
5. Participants who can understand and follow the research process, voluntarily participate, and sign an informed consent form (informed consent is voluntarily signed by the person or legal representative).

Exclusion Criteria:

1. Known to be allergic to research drugs or similar ingredients, or materials used in imaging studies;
2. Weight >120kg or <45kg;
3. The timing of stroke symptoms is not known;
4. mRS score before stroke≥ 2 points;
5. NIHSS score 1a (level of consciousness) ≥ 2 points during screening;
6. Patients with intracerebral hemorrhage history;
7. CT/MRI imaging examination shows signs of intracranial hemorrhage or suspected subarachnoid hemorrhage despite CT/MRI imaging findings do not show abnormalities;
8. Severe cerebral trauma or stroke history or other severe traumas within 3 months;
9. Assessment of Intracranial tumor, arteriovenous malformation and aneurysm before admission;
10. Intracranial surgery, intraspinal surgery or other major surgeries within 3 months (based on the assessment of the investigators);
11. Patients with gastrointestinal or urinary system hemorrhage in recent 3 weeks;
12. Active visceral hemorrhage;
13. Assessment or with history of aortic arch dissection before admission;
14. Arterial puncture in 1 week which can not be oppressed;
15. Subjects who have an acute bleeding tendency, including but not limited to：1) a platelet count of less than 100 × 109 / L；2) application of low molecular heparin within 24 hours before onset ; 3) Using of thrombin inhibitors or factor Xa inhibitor within 48 hours before onset ; 4) application of oral anticoagulant drugs and with an INR > 1.7 or PT>15s;
16. Hypertension remains uncontrolled after active antihypertensive therapy, uncontrolled hypertension refers to a systolic blood pressure >185 mmHg and/or a diastolic blood pressure >110 mmHg;
17. Blood glucose <50 mg/dl (equivalent to 2.78mmol/L) or >400 mg/dl (equivalent to 22.2mmol/L);
18. Imaging (CT or MRI)shows large area cerebral infarction;
19. Severe liver damage, including liver failure, cirrhosis, portal hypertension (esophageal varices), and active hepatitis;
20. Bacterial endocarditis or pericarditis, acute pancreatitis at admission;
21. With history of gastrointestinal ulcers, esophageal varices, aneurysms, or arterial / venous malformations within 3 months before admission;
22. Patients who are unable to cooperate or are unwilling to cooperate with epileptic seizures, or other mental illnesses during stroke episodes;
23. Patients who are ready to go or have undergone endovascular treatment;
24. The restricted drug specified in the protocol or any drug that may interfere with the test results must be ingested or desired to continue to be ingested;
25. An expected survival time of no more than 1 year due to other diseases;
26. Patients who are participating in other trials or have participated in other trials within 30 days before randomization;
27. Pregnancy or lactation, or women who have a positive pregnancy test result;
28. The subject who is unsuitable for this study in the opinion of the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1412 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Functional handicap | on the 90th day after treatment
  Proportion of patients achieving a Modified Rankin Scale score of 0 to 1 on the 90th day after treatment.
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0-5. A separate category of 6 is usually added for patients who expire. The higher the score, the more severe the stroke.

SECONDARY OUTCOMES:
Proportion of Neurological Improvement | at 24hours and the 7th day after treatment
  The proportion of subjects with NIHSS score ≤1 or the decrease of 4 points or more from the baseline at 24 hours and the 7th day after treatment.
  The National Institutes of Health Stroke Scale (NIHSS) is a 11-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on level of consciousness, eye movements, integrity of visual fields, facial movements,arm and leg muscle strength, sensation, coordination, language,speech and neglect. Each impairment is scored on an ordinal scale ranging from 0 to 2, 0 to 3, or 0 to 4. Item scores are summed to a total score ranging from 0 to 42 (the higher the score, the more severe the stroke).
Proportion of Long-term Improvement | on the 90th day after treatment
  Proportion of patients achieving a mRS of 0 to 2 on the 90th day after treatment.
Ordinary distribution of mRS scores | on the 90th day after treatment
  Ordinary distribution of mRS scores on the 90th day after treatment.
Barthel Index score | on the 90th day after treatment
  Proportion of patients achieving a Barthel Index score ≥95 on the 90th day after treatment.
  The Barthel Index of Activities of Daily Living (ADLs) measures functional disability by quantifying patient performance in 10 activities of daily life. These activities can be grouped according to self-care (feeding, grooming, bathing, dressing, bowel and bladder care, and toilet use) and mobility (ambulation, transfers, and stair climbing). 5-point increments are used in scoring, with a maximal score of 100 indicating that a patient is fully independent in physical functioning, and a lowest score of 0 representing a totally dependent bed-ridden state.

OTHER OUTCOMES:
Proportion of subjects died of all cause | within 7 days and 90 days after treatment
  All-cause mortality within 7 days and 90 days after treatment.
Percentage of subjects with symptomatic intracranial hemorrhage (sICH) | SITS criteria: within 36 hours after treatment; ECASS III criteria: within 36 hours and 7 days after treatment
  sICH definition: 1. SITS criteria: local or remote parenchymal hematoma type 2 on the imaging scan obtained within 36 hours after treatment, plus neurologic deterioration, as indicated by a score on the NIHSS that was higher by 4 points or more than the baseline value or the lowest value between baseline and 24 hours, or hemorrhage leading to death. 2. The ECASS III criteria：any hemorrhage with neurologic deterioration, as indicated by an NIHSS score that was higher by 4 points or more than the value at baseline or the lowest value in the first 7 days , or any hemorrhage leading to death. In addition, the hemorrhage must have been identified as the predominant cause of the neurologic deterioration (This study will be evaluated and recorded according to the above two standards).
Proportion of subjects with major hemorrhage and clinically relevant non-major hemorrhage（ISTH criteria） | within 90 days after treatment
  ISTH：International Society of Thrombosis and Hemostasis.
The Proportion of subjects with AE、SAE | within 90 days after treatment
  The Proportion of subjects with AE、SAE within 90 days after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Principal Investigator — Beijing Tiantan Hospital
Locations (78):
- China (78):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Chongqing Emergency Medical Center, Chongqing, Chongqing Municipality
  - Gaozhou People's Hospital, Gaozhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Yue Bei People's Hospital, Shaoguan, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hebei Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine, Cangzhou, Hebei
  - Handan Central Hospital, Handan, Hebei
  - Hengshui People's Hospital, Hengshui, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan Workers'Hospital, Tangshan, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Daqing People's Hospital, Daqing, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Third Affiliated Hospital of Qiqihar Medical College, Qiqihar, Heilongjiang
  - Anyang People's Hospital, Anyang, Henan
  - Jiaozuo People's Hospital, Jiaozuo, Henan
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyan, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Luoyang Central Hospital, Luoyang, Henan
  - Nanyang Nanshi Hospital, Nanyang, Henan
  - Nanyang Second People's Hospital, Nanyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - Zhengzhou People's Hospital, Zhengzhou, Henan
  - Zhumadian Central Hospital, Zhumadian, Henan
  - Wuhan Fourth Hospital (Wuhan Puai Hospital, Wuhan Orthopaedic Hospital), Wuhan, Hubei
  - The First Affiliated Hospital of Nanhua University, Hengyang, Hunan
  - Yiyang Central Hospital, Yiyang, Hunan
  - Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology, Baotou, Inner Mongolia
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Huai'an Second People's Hospital, Huai'an, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Yichun People's Hospital, Yichun, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - Jilin People's Hospital, Jilin, Jilin
  - Meihekou Central Hospital, Meihekou, Jilin
  - Jilin Guowen Hospital, Siping, Jilin
  - Tonghua Central Hospital, Tonghua, Jilin
  - Fukuang General Hospital of Liaoning Health Industry Group, Fushun, Liaoning
  - First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - PLA Northern Theater Command General Hospital, Shenyang, Liaoning
  - Shenyang First People's Hospital, Shenyang, Liaoning
  - Central Hospital Affiliated to Shenyang Medical College, Shenyang, Liaoning
  - Dezhou People's Hospital, Dezhou, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Qianfo Mountain Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical College, Jining, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Tai'an Central Hospital, Tai’an, Shandong
  - Weifang Hospital of Traditional Chinese Medicine, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai Pudong Hospital, Shanghai, Shanghai Municipality
  - General Hospital of Tongmei Group, Datong, Shanxi
  - Yan'an University Xianyang Hospital, Xianyang, Shanxi
  - Xi'an Daxing Hospital, Xi’an, Shanxi
  - Xi'an High-tech Hospital 204 Hospital, Xi’an, Shanxi
  - Zigong First People's Hospital, Zigong, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - First People's Hospital of Kashgar Region, Kashgar, Xinjiang
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Jiaxing First Hospital, Jiaxing, Zhejiang
  - Taizhou First People's Hospital, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Feng B, Gu HQ, Li Z, Wang Y, Zhao X, Li S, Wang Y. Outcomes of Time to Treatment With Reteplase for Acute Ischemic Stroke: The RAISE Trial Subgroup. JACC Asia. 2025 Apr;5(4):584-592. doi: 10.1016/j.jacasi.2024.12.010. Epub 2025 Feb 11. PMID 40180551
- [Derived] Li S, Gu HQ, Li H, Wang X, Jin A, Guo S, Lu G, Che F, Wang W, Wei Y, Wang Y, Li Z, Meng X, Zhao X, Liu L, Wang Y; RAISE Investigators. Reteplase versus Alteplase for Acute Ischemic Stroke. N Engl J Med. 2024 Jun 27;390(24):2264-2273. doi: 10.1056/NEJMoa2400314. Epub 2024 Jun 14. PMID 38884332
- [Derived] Li S, Gu HQ, Dai H, Lu G, Wang Y. Reteplase versus alteplase for acute ischaemic stroke within 4.5 hours (RAISE): rationale and design of a multicentre, prospective, randomised, open-label, blinded-endpoint, controlled phase 3 non-inferiority trial. Stroke Vasc Neurol. 2024 Nov 5;9(5):568-573. doi: 10.1136/svn-2023-003035. PMID 38286482